CLINICAL TRIAL: NCT03029572
Title: Micro-nutritional Status and Gut Microbiota in Morbidly Obese Patients Before and After Gastric Bypass With and Without Micro-nutritional Supplementation
Brief Title: Micro-nutritional Status and Gut Microbiota in Morbidly Obese Patients Before and After Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Zoltan Pataky, Deputy Head, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-005
Record Dates: First submitted 2017-01-14; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard diet (Active Comparator): Standard healthy diet after RYGB surgery
  Interventions: Procedure: Bariatric surgery
- Micro-nutriments' supplementation (Experimental): Healthy diet and probiotics, minerals, aminoacids, omega-3 acids vitamin and mineral supplementation after RYGB surgery
  Interventions: Drug: Diet supplementation; Procedure: Bariatric surgery

INTERVENTIONS:
Drug: Diet supplementation — Micronutriment supplementation therapy
  Arms: Micro-nutriments' supplementation
Procedure: Bariatric surgery — Roux-en-Y gastric bypass provided in both arms.

SUMMARY:
An intervention study design in 90 obese patients will be used. Nutritional, metabolic and psychological status as well as gut microbiota will be evaluated before gastric bypass and 6 months post surgery. During this period of 6 months, all patients will receive a specific diet according to recommendation with regard to bariatric surgery.

Subjects will be than randomized in 2 sub-groups:

A. patients receiving a standard healthy diet without micro-nutriments' supplementation; B. patients receiving a healthy diet and probiotics, minerals, aminoacids, omega-3 acids vitamin and mineral supplementation

DETAILED DESCRIPTION:
The primary aim of the study is to analyse the micro-nutritional status in morbidly obese patients before and 6 months after bariatric surgery (Roux-en-Y gastric bypass, RYGB). The secondary outcome will be the impact of 6 months probiotics, minerals, aminoacids, omega-3 acids and vitamin supplementation on microbiota, metabolic and psychological parameters 12 months post-RYGB.

An intervention study in 90 obese patients (BMI>40 kg/m2) will be used. Nutritional, metabolic and psychological status as well as gut microbiota will be evaluated before gastric bypass and 6 months post RYGB. During this period of 6 months, all patients will receive a specific diet according to recommendation with regard to RYGB.

Subjects will be than randomized in 2 sub-groups:

A. patients receiving a standard healthy diet without micro-nutriments' supplementation; B. patients receiving a healthy diet and probiotics, minerals, aminoacids, omega-3 acids vitamin and mineral supplementation Healthy diet will be defined as follow: 9-15% of proteins, 50-55% of carbohydrates and 30-35% lipids (25% saturated fat, 50% mono-unsaturated fat and 25% poly-unsaturated fat).

The following parameters will be analysed before RYGB and 6 months and 12 months post RYGB, respectively:

* Nutritional status with oxidative stress parameters (Vitamins A and E, Selenium, Zinc, Copper, Glutathione peroxidise, Superoxide dismutase and Iron)
* Metabolic parameters (Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides, fasting glucose and insulin, CRP)
* Fatty acids (linoleic acid, alpha-linoleic acid (ALA), eicosapentaenoic acid (EPA), and docosahexaenoic acid (DHA)
* Gut microbiota
* Psychological status (anxiety, depression and quality of life as evaluated by validated questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Obesity BMI>40 kg/m2

Exclusion Criteria:

* Antidepressant treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Vitamins A levels | Change from Baseline at 6-months and 12-months post-RYGB
Vitamin E levels | Change from Baseline at 6-months and 12-months post-RYGB
Selenium levels | Change from Baseline at 6-months and 12-months post-RYGB
Zinc levels | Change from Baseline at 6-months and 12-months post-RYGB
Copper levels | Change from Baseline at 6-months and 12-months post-RYGB
Glutathione peroxidise | Change from Baseline at 6-months and 12-months post-RYGB
Superoxide dismutase | Change from Baseline at 6-months and 12-months post-RYGB
Iron levels | Change from Baseline at 6-months and 12-months post-RYGB

SECONDARY OUTCOMES:
Total cholesterol | 6-months and 12-months post-RYGB
LDL-cholesterol | 6-months and 12-months post-RYGB
HDL-cholesterol | 6-months and 12-months post-RYGB
Triglycerides | 6-months and 12-months post-RYGB
Fasting glucose | 6-months and 12-months post-RYGB
Fasting insulin | 6-months and 12-months post-RYGB
C-Reactive Protein | 6-months and 12-months post-RYGB
Linoleic acid | 6-months and 12-months post-RYGB
Alpha-linoleic acid (ALA) | 6-months and 12-months post-RYGB
Eicosapentaenoic acid (EPA) | 6-months and 12-months post-RYGB
Docosahexaenoic acid (DHA) | 6-months and 12-months post-RYGB
Gut microbiota modifications (sequencing the V4 region of 16S rDNA) | 6-months and 12-months post-RYGB
Anxiety (questionnaire HAD) | 6-months and 12-months post-RYGB
Depression (questionnaire HAD) | 6-months and 12-months post-RYGB
Quality of life (questionnaire IWQOL) | 6-months and 12-months post-RYGB

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No